CLINICAL TRIAL: NCT01264185
Title: Preparing for International Prevention Trials Involving HIV-Infected Individuals in Care Settings
Acronym: HPTN063
Status: Completed | Type: Observational
Sponsor: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Other Study IDs: HPTN 063
Record Dates: First submitted 2010-12-14; First posted 2010-12-21 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, genital fluids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asia--Thailand; S. America--Brazil
- Africa--Zambia

SUMMARY:
The purpose of this study is to conduct preparatory research needed to design a behavioral intervention to decrease sexual transmission risk behaviors in HIV-infected individuals in care and to determine whether a similar intervention structure can be used across various sexual risk groups and cultural settings.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age (Note: Pregnant and breast feeding women are allowed to enroll into the study)
* Documented evidence of HIV infection (HIV diagnosis performed outside of the trial is acceptable so long as local/country guidelines were followed in the testing)
* Receiving HIV/AIDS care (defined as at least two visits within 9 months of enrollment) in a formal health care setting (clinic or hospital)
* Reported history of sexual risk behavior in the previous 12 months, including: acquisition of a sexually transmitted infection, vaginal or anal intercourse without a condom, difficulty negotiating condom use, or non-disclosure of HIV status to an HIV-uninfected partner or partner of unknown HIV serostatus.
* NOTE: For the MSM population, we will enroll men who have sex with men, regardless of whether or not they also have sex with women

Exclusion Criteria:

* Anyone currently enrolled in another study that involves protocolized HIV risk reduction counseling (e.g. ACTG 5175 or HPTN 052) or any other prevention study
* Anyone having unprotected (i.e. without a condom) sex for the expressed purpose of conceiving
* Planning to relocate out of the area in the next year
* Any condition that, in the opinion of the Investigator of Record or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asia (Thailand) and South America (Brazil)
  * 100 heterosexual men,
  * 100 heterosexual women,
  * 100 Men having sex with men (MSM), and
  * ~40 community members and stakeholders
  Africa (Zambia)
  * 100 heterosexual men,
  * 100 heterosexual women,
  * ~40 community members and stakeholders
Sampling Method: Non-Probability Sample
Enrollment: 751 (Actual)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Establish baseline rates of sexual HIV transmission risk | 1 year
  To establish baseline rates of sexual HIV transmission risk behavior in high risk HIV-infected individuals, and to observe the rates and patterns of behavior change over time
Structure and content of a behavioral intervention for individuals with HIV | 1 year
  To gather formative data on the potential structure and content of a behavioral intervention for individuals with HIV in care in international settings and to determine the best, culturally appropriate model for the intervention that will link prevention to care for HIV-infected individuals.
Identify psychosocial and sociodemographic correlates of sexual risk-taking | 1 year
  To examine potential psychosocial and sociodemographic correlates of sexual risk-taking in these individuals in order to help shape the content of an individualized behavioral intervention

SECONDARY OUTCOMES:
Determine sexually transmitted infection(STI)prevalence and incidence | 1 year
  Evaluate STI prevalence and incidence and investigate whether these biomarkers may be used to corroborate self-reported sexual behavior associated with potential transmission risks

CONTACTS AND LOCATIONS:
Overall Officials: Steve Safren, PhD, Study Chair — Fenway Community Health Center; Ken Mayer, MD, Study Chair — Fenway Community Health Center; Stewart Reid, MD, MPH, Principal Investigator — Centre for Infectious Disease Research in Zambia (CIDRZ); Ruth Friedman, MD, Principal Investigator — Instituto de Pesquisa Clincia Evandro Chagas (IPEC) Clinical Research Site (CRS); Kriengkrai Srithanaviboonchai, MD, MPH, Principal Investigator — Chiang Mai University AIDS CRS
Locations (3):
- Instituto de Pesquisa Clinicaq Evandro Chagas CRS, Manguinhos, Rio de Janeiro, Brazil
- Chiang Mai University AIDS CRS, Chiang Mai, Thailand
- Matero Reference Clinic, Lusaka, Zambia